CLINICAL TRIAL: NCT06943976
Title: The Value of PROMs in Children With Hearing Loss: Patients', Parents' and Healthcare Professionals' Perspectives
Brief Title: How Parents, Children, and Clinicians Experience Digital Health Tools in Pediatric Audiology
Status: Not yet recruiting | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Christina Batthyany, Resident and PhD Candidate in Otorhinolaryngology - Head and Neck Surgery, Erasmus Medical Center
Other Study IDs: 13562
Record Dates: First submitted 2025-04-17; First posted 2025-04-25 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Hearing Loss, Bilateral or Unilateral
Keywords: Hearing Loss; Quality of Life; PROMs; PREMs; Children; Digital Health Care
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to understand how children with hearing loss, their parents, and health care providers experience digital health questionnaires that are completed before audiology follow-up appointments. The study focuses on children and adolescents (aged 7-18 years old) with hearing loss, and their parents, visiting the Audiology outpatient clinic of the Erasmus MC Sophia Children's Hospital.

The main questions it aims to answer are:

* How do parents, children, and clinicians experience digital questionnaires like the HEAR-QL before an audiology visit?
* Do these digital tools help improve communication and preparation for the appointment?

Participants will:

* Be invited to complete a short feedback questionnaire about their experience with digital tools
* Share their views on how helpful or relevant the questionnaires were
* Health care providers will also give feedback on how they use and interpret the responses in clinical care

DETAILED DESCRIPTION:
This observational study evaluates the experiences of children with hearing loss, their parents or caregivers, and audiology health care providers with digital health questionnaires that are completed before pediatric audiology follow-up visits. The study is conducted at the Audiology outpatient clinic of the Erasmus MC Sophia Children's Hospital in Rotterdam, the Netherlands.

As part of routine clinical care, families receive electronic patient-reported outcome measures (PROMs) prior to their appointment, including the Dutch versions of the HEAR-QL questionnaire. These questionnaires are designed to gather insights into the child's hearing-related quality of life and relevant experiences related to hearing care.

Participants in this study include children and adolescents (ages 7-18 years) with unilateral or bilateral hearing loss, their caregivers, and health care professionals (audiologists, speech language pathologists and/or ENT specialists). All participants are invited to provide feedback on the digital questionnaires via brief evaluation surveys (PREMs). This information is collected anonymously and used to understand the usability, relevance, and clinical value of the tools from both the patient and provider perspectives.

Registry-related procedures and quality factors:

* Quality assurance plan: All data are collected using a secure digital platform. Data entry is automated via survey completion, reducing the risk of manual input errors. Registry procedures follow institutional data management standards.
* Data checks and validation: Built-in logic and range checks are applied within the digital survey software to prevent incomplete or inconsistent responses.
* Source data verification: No source data verification is applied, as this study does not use patient medical records beyond the standard demographic and audiological information collected with informed consent.
* Data dictionary: A standardized variable list is maintained, including definitions, coding schemes, and units of measurement. The HEAR-QL scoring methodology is applied as per published validation guidelines.
* Standard Operating Procedures (SOPs): SOPs exist for patient approach, informed consent, survey distribution, data storage, and privacy protection. All procedures align with institutional review board approvals.
* Sample size: The study aims to include a minimum of 50 families (about 80 respondents) over a 4-month period, which is sufficient for descriptive and exploratory analyses of user experience outcomes.
* Missing data: Missing data is not expected, as all questions in the digital questionnaires are required fields. The system prevents submission of incomplete surveys. Therefore, no item-level missingness or imputation procedures are applicable.
* Statistical analysis plan: Quantitative survey responses will be summarized using descriptive statistics (e.g., means, medians, proportions). Associations between user experience scores and patient characteristics (e.g., age, hearing device type) may be explored using nonparametric tests or regression analyses as appropriate. Qualitative comments from participants will be grouped thematically.

This study aims to contribute to the growing body of knowledge on patient and provider experiences with digital health tools in pediatric audiology. Results may inform future implementation and optimization of PROMs in routine hearing care.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents, aged 7-18 years old, with rehabilitated unilateral or bilateral hearing loss, attending the Audiology outpatient clinic of the Erasmus MC Sophia Children's Hospital in Rotterdam, the Netherlands
* The corresponding parents or caregivers of these pediatric patients
* Audiologists or other health care providers who systematically use the PROMs during patient interactions at the same Audiology outpatient clinic.

Exclusion Criteria:

* Children or adolescents who are unable to complete the questionnaire, even with support in reading and understanding the items provided by their parents or caregivers.

Ages: 7 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants will be selected from the population of children and adolescents aged 7 to 18 years with unilateral or bilateral hearing loss who attend the Audiology outpatient clinic of Erasmus MC Sophia Children's Hospital in Rotterdam, the Netherlands. Their parents or primary caregivers will also be invited to participate. Additionally, audiologists and other health care professionals working at the same clinic and using patient-reported outcome measures (PROMs) in routine care will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Experience with digital health questionnaires | Within 3 months after the audiology appointment
  Experience scores from a custom feedback survey completed by parents/caregivers and children aged 7-18 years, evaluating clarity, relevance, and burden of digital questionnaires.

SECONDARY OUTCOMES:
Clinician-perceived utility of digital questionnaires | Within the time frame of the patient enrollment
  Ratings from audiology/health care staff on the usefulness of digital patient-reported outcome measures (PROMs) in preparing for or guiding the consultation.